CLINICAL TRIAL: NCT00979979
Title: Clinical Performance of Abbott RealTime HCV Genotype II Test
Brief Title: Clinical Performance of Abbott RealTime Hepatitis C Virus (HCV) Genotype II Test
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Abbott Diagnostics Division (Industry); National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200906047D
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Genotype; Realtime PCR
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Patient stored serum with detectable HCV RNA levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV patients: HCV patients with detectable viremia; all sera are tested both by Abbott RealTime HCV genotype II test and by direct HCV sequencing both at 5'UTR and NS5B
- Non-HCV patients: Patient without evidence of HCV infection (negative both for anti-HCV and HCV RNA); all sera are both tested by Abbott RealTime HCV genotype II test and by direct HCV sequencing at 5'UTR and NS5B

SUMMARY:
Hepatitis C virus (HCV) infection, a leading cause of cirrhosis, hepatocellular carcinoma (HCC) and liver transplantation, affects approximately 170 million individuals worldwide. Combination of peginterferon plus ribavirin therapy has become the current standard of care for chronic hepatitis C (CHC) patients, with an overall sustained virologic response (SVR) rate of 54-63% and more favorable response rates in patients with genotype 2/3 infection than those with genotype 1/4 infection. Therefore, accurate pre-treatment HCV genotype evaluation is of paramount importance to facilitate individualized therapy in the era of response guide therapy and specific-targeted antiviral therapy for HCV (STAT-C).

Currently, direct HCV genetic sequencing for both the 5' untranslated terminal region (5'UTR) and non-structural 5B (NS5B) regions with subsequent phylogenetic tree analysis is considered the gold standard for determining HCV genotype and subtype. However, it is time-consuming and need special laboratory settings. Several commercial available reverse hybridization with type-specific probing assay (Inno-LiPA II) or simplified direct sequencing of the 5'UTR region were used to replace the two region sequencing method (Trugene HCV 5' NC genotyping kit). Nonetheless, data on the overall diagnostic accuracy varied.

The Abbott RealTime HCV Genotype II is an in vitro reverse transcription-polymerase chain reaction (RT-PCR) assay for determining the genotype(s) of HCV in plasma and serum from HCV-infected individuals. Based on genetic similarity, HCV has been classified into six major genotypes (1-6) and numerous subtypes. HCV genotype is predictive of the response of HCV-infected patients to peginterferon plus ribavirin combination therapy. The Abbott RealTime HCV Genotype II assay uses the Abbott m2000sp instrument for processing samples and the Abbott m2000rt instrument for amplification and detection. Furthermore, the Abbott m2000sp provides automated sample transfer and reaction assembly of the assay reagents in the Abbott 96-Well Optical Reaction Plate.

The investigators aimed to evaluate the overall diagnostic accuracy of the currently available commercial HCV genotype kits (Abbott RealTime HCV Genotype II) by using 5'UTR and NS5A gene amplification and direct sequencing as the gold standard.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection, a leading cause of cirrhosis, hepatocellular carcinoma (HCC) and liver transplantation, affects approximately 170 million individuals worldwide. Therefore, prevention of HCV transmission and early intervention of HCV infection are urgently needed to reduce or halt the liver-related morbidity and mortality. Combination of peginterferon plus ribavirin therapy has become the current standard of care for chronic hepatitis C (CHC) patients, with an overall sustained virologic response (SVR) rate of 54-63% and more favorable response rates in patients with genotype 2/3 infection than those with genotype 1/4 infection. Therefore, accurate pre-treatment HCV genotype evaluation is of paramount importance to facilitate individualized therapy in the era of response guide therapy and specific-targeted antiviral therapy for HCV (STAT-C).

Currently, direct HCV genetic sequencing for both the 5' untranslated terminal region (5'UTR) and non-structural 5B (NS5B) regions with subsequent phylogenetic tree analysis is considered the gold standard for determining HCV genotype and subtype. However, it is time-consuming and need special laboratory settings. Several commercial available reverse hybridization with type-specific probing assay (Inno-LiPA II) or simplified direct sequencing of the 5'UTR region were used to replace the two region sequencing method (Trugene HCV 5' NC genotyping kit). Nonetheless, data on the overall diagnostic accuracy varied.

The Abbott RealTime HCV Genotype II is an in vitro reverse transcription-polymerase chain reaction (RT-PCR) assay for determining the genotype(s) of HCV in plasma and serum from HCV-infected individuals. Based on genetic similarity, HCV has been classified into six major genotypes (1-6) and numerous subtypes. HCV genotype is predictive of the response of HCV-infected patients to peginterferon plus ribavirin combination therapy. The Abbott RealTime HCV Genotype II assay uses the Abbott m2000sp instrument for processing samples and the Abbott m2000rt instrument for amplification and detection. Furthermore, the Abbott m2000sp provides automated sample transfer and reaction assembly of the assay reagents in the Abbott 96-Well Optical Reaction Plate.

The investigators aimed to evaluate the overall diagnostic accuracy of the currently available commercial HCV genotype kits (Abbott RealTime HCV Genotype II) by using 5'UTR and NS5A gene amplification and direct sequencing as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* HCV patients with both positive for anti-HCV and HCV RNA (Cobas Taqman, Roche Diagnostics, LOQ:25 IU/mL and LOD:10 IU/mL)
* Patients with signed informed consent

Exclusion Criteria:

* Patients without signed informed consent
* HCV patients without detectable HCV RNA (Cobas Taqman, Roche Diagnostics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 255 HCV patients both positive for anti-HCV and HCV RNA and 18 patients without ant-HCV and HCV RNA; all 255 patients were tested for Abbott RealTime genotype II test and direct HCV sequencing at 5'UTR and NS5B for the sensitivity, specificity, and the overall diagnostic accuracy.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2009-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for HCV genotype testing | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — National Taiwan University Hospital; Jia-Horng Kao, MD, PhD, Study Director — National Taiwan University Hospital; Chun-Jen Liu, MD, PhD, Principal Investigator — National Taiwan University Hospital; Cheng-Chao Liang, MD, BS, Principal Investigator — Far Eastern Memorial Hospital; Chih-Lin Lin, MD, BS, Principal Investigator — Taipei Municipal Hospital, Ren-Ai Branch; Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (4):
- Taiwan (4):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Far Eastern Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Hospital, Ren-Ai Branch, Taipei

REFERENCES:
- [Derived] Liu CH, Liang CC, Liu CJ, Lin CL, Su TH, Yang HC, Chen PJ, Chen DS, Kao JH. Comparison of Abbott RealTime HCV Genotype II with Versant line probe assay 2.0 for hepatitis C virus genotyping. J Clin Microbiol. 2015 May;53(5):1754-7. doi: 10.1128/JCM.03548-14. Epub 2015 Mar 4. PMID 25740780